CLINICAL TRIAL: NCT03190252
Title: Biokemiska förändringar Vid förhöjt Partialtryck för Syrgas
Brief Title: Inflammatory and Cerebrospinal Biochemical Markers in Blood After Trimix Diving
Acronym: TriMix17-18
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Göteborg University (Other); Swedish Armed Forces Diving and Naval Medicine Centre (Other); KTH Royal Institute of Technology (Other)
Responsible Party: Principal Investigator, Anders Rosén, MD PhD student, Sahlgrenska University Hospital
Other Study IDs: EPN 292-17
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Diving Medicine; Inflammation; Central Nervous System Injury
Keywords: Diving medicine; Inflammation; Central nervous system injury; Trimix; Decompression sickness; Venous gas emboli
MeSH Terms: conditions — Inflammation; Decompression Sickness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, Serum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trimix: Exposure to ambient pressure of maximum 11 ATA breathing Trimix. Exposure to oxygen partial pressure of 130 kPa breathing Trimix.
  Interventions: Other: Exposure to oxygen partial pressure of 130 kPa; Other: Exposure to ambient pressure of maximum 11 ATA

INTERVENTIONS:
Other: Exposure to oxygen partial pressure of 130 kPa — Open sea diving to a maximum depth of 100 msw while breathing Trimix.
Other: Exposure to ambient pressure of maximum 11 ATA — Open sea diving to a maximum depth of 100 msw while breathing Trimix.

SUMMARY:
Research hypothesis

* Diving to depths up to 90msw with an oxygen partial pressure of 130kPa in the breathing gas will affect the central nervous system.
* Diving to depths up to 90msw with an oxygen partial pressure of 130kPa in the breathing gas will induce inflammatory changes.

Objectives:

* To investigate the presence of cerebrospinal biochemical markers in blood after diving to depths up to 90msw with an oxygen partial pressure of 130kPa in the breathing gas.
* To investigate the presence of inflammatory markers in blood after diving to depths up to 90msw with an oxygen partial pressure of 130kPa in the breathing gas.
* To investigate the presence of venous gas emboli (VGE) in blood after diving to depths up to 90msw with an oxygen partial pressure of 130kPa in the breathing gas.

DETAILED DESCRIPTION:
When diving with compressed air as breathing gas, a continuous accumulation of nitrogen will take place in the body. The total uptake of nitrogen by the tissues is dependent on the duration and depth of the performed dive. Decompression at the end of a dive can cause accumulated nitrogen to form intravascular bubbles.

Furthermore, at depths greater than 30 meters seawater (msw) the elevated partial pressure of nitrogen in the breathing gas will exert a direct effect on the nervous system. This is known as nitrogen narcosis and can cause altered cognitive function, confusion, behavioural disturbance and altered level of consciousness. The effect of nitrogen narcosis gets more pronounced with increasing diving depth. To avert nitrogen narcosis it is common to reduce the amount of nitrogen in the breathing gas being used. At the same time the amount of oxygen must also be reduced, as partial pressures of oxygen above 1,6kPa could induce seizures. Usually a breathing gas mixture containing helium, nitrogen and oxygen (TriMix) is used.

It has long been considered that decompression sickness (DCS) is caused by bubble formation when dissolved nitrogen at the end of diving comes out of solution. Doppler ultrasound techniques have shown that intravascular gas bubbles could exist even after uneventful dives. Therefore, additional pathophysiological factors must be sought.

There is evidence of an increased inflammatory activity in blood after diving. Signs of neutrophil activation is a common finding. It is not known if hyperbaric exposure in itself is enough to elicit these biochemical changes or if the presence of intravascular nitrogen bubbles is needed.

Studies have shown that biochemical markers of central nervous system (CNS) injury can be detected in blood samples obtained from patients with DCS, metabolic and neurologic disease, during cardiac surgery and after traumatic brain injuries. Such markers can also be seen in blood after sport activities like boxing and breath hold diving. If biochemical markers of CNS injury will be present in blood after hyperbaric exposure is not known.

The Swedish armed forces (SwAF) Diving and Naval Medicine Center (DNC) is responsible for education and training of divers for SwAF. The centre is also responsible for research and development and conduct tests for diving medicine, and tests of underwater equipment.

SwAF DNC will during 2017 and 2018 be responsible for naval dive training including deep dives (up to 90 msw) using TriMix as breathing gas. The partial pressure of oxygen will be kept at 130kPa. The study "Inflammatory and cerebrospinal biochemical markers in blood after TriMix diving - an observational controlled study" will be followed out during these tests. It entails venous blood sampling and cardiac ultrasound.

This is a prospective, controlled observational study (see addendum 08/03/19 below). The study aims to involve at least 16 study subjects. Half of the subjects (at least 8 persons), named the intervention group, dive to depths up to 90msw with an oxygen partial pressure of 130kPa in the TriMix breathing gas. Half of the subjects (at least 8 persons), named the control group, do not dive. The dives are part of the Swedish navy´s training programme for TriMix diving.

Blood samples are obtained from the intervention group before and after diving (two tubes and about 8mL of blood each time, in total 16mL of blood). If possible, a third blood sample are taken about 24 hours after the first sample. Blood samples are obtained from the control group at the same time points as from the intervention group.

Immmediately after diving, cardiac ultrasound will be used to assess presence and duration of VGE in the intervention group.

Signs of DCS will be actively sought.

Addendum 08/03/19: A control group containing non-diving military divers was initially planned. However, difficulties in subject recruitment meant that an appropriate control group could not be formed. It was performed as an observational study without controls.

ELIGIBILITY:
Inclusion Criteria:

- Military diver or individual approved by the Swedish navy to dive or perform work in hyperbaric environments

Exclusion Criteria:

- As this is a highly selected population there is no exclusion criteria

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Military divers and individuals approved by the Swedish navy to dive or perform work in hyperbaric environment.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Concentration of cerebrospinal and inflammatory biochemical markers in blood | Three months
  E.g. GFAP, Tau, NfL, JCHL-1, VCAM-1, ICAM-1

SECONDARY OUTCOMES:
Presence of Venous Gas Emboli (VGE) | Five days
  Kisman-Masurel grading
Decompression Sickness (DCS) | Five days
  Clinical diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Zetterberg, PhD, Study Director — Göteborg University
Locations (1):
- Gothenburg University, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No